CLINICAL TRIAL: NCT00151242
Title: Randomized Phase II/III-Study on All-Trans Retinoic Acid in Combination With Induction and Consolidation Therapy as Well as Pegfilgrastim After Consolidation Therapy in Younger Patients With Newly Diagnosed Acute Myeloid Leukemia
Brief Title: Study on All-Trans Retinoic Acid, Induction and Consolidation Therapy, and Pegfilgrastim After Consolidation Therapy in Younger Patients With Newly Diagnosed Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Prof. Dr. Richard Schlenk, PD Dr., University of Ulm
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMLSG07-04
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; Idarubicin; Etoposide; Tretinoin; pegfilgrastim

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Cytarabine; Drug: Idarubicin; Drug: Etoposide; Drug: Pegfilgrastim
- 2 (Experimental)
  Interventions: Drug: Cytarabine; Drug: Idarubicin; Drug: Etoposide; Drug: All-trans retinoic acid; Drug: Pegfilgrastim

INTERVENTIONS:
Drug: Cytarabine — 100mg/m² kont. i.v. day 1-7 (induction therapy) 3g/m² 2x/die i.v. day 1,3,5 or day 1,2,3
Drug: Idarubicin — 12mg/m² i.v. day 1,3,5 (first induction cycle) 12mg/m² i.v. Tag 1,3 (second induction cycle)
Drug: Etoposide — 100mg/m² i.v. day 1-3 (induction therapy)
Drug: All-trans retinoic acid — 45mg/m² p.o. day 6-8 (induction therapy) 15mg/m² p.o. day 9-21 (induction therapy) 15mg/m² p.o. day 6-21 (consolidation therapy)
  Arms: 2
Drug: Pegfilgrastim — 6mg s.c day 10 (cohort 1), 6mg s.c. day 8 (cohort 2)
  Other Names: Neulasta

SUMMARY:
This trial is a study on all-trans retinoic acid in combination with induction and consolidation therapy as well as pegfilgrastim after consolidation therapy in younger patients with newly diagnosed acute myeloid leukemia (AML).

DETAILED DESCRIPTION:
First Induction Therapy:

* Cytarabine 100 mg/m² cont. i.v. days 1-7
* Idarubicin 12 mg/m² i.v. days 1,3,5
* Etoposide 100 mg/m² i.v. days 1-3
* ± ATRA 45 mg/m² p.o. days 6-8
* ATRA 15 mg/m² p.o. days 9-21

Second Induction Therapy:

* Cytarabine 100 mg/m² cont. i.v. days 1-7
* Idarubicin 12 mg/m² i.v. days 1 and 3
* Etoposide 100 mg/m² i.v. days 1-3
* ± ATRA 45 mg/m² p.o. days 6-8
* ATRA 15 mg/m² p.o. days 9-21

Consolidation Therapy:

cohort 1 (<= ID 336)

* Cytarabine 3 g/m² 2x/die i.v. Tag 1,3,5
* ± ATRA 15 mg/m² p.o. Tag 6-21
* Pegfilgrastim 6 mg s.c day 10

cohort 2 (> ID 336)

* Cytarabine 3 g/m² 2x/die i.v. Tag 1,2,3
* ± ATRA 15 mg/m² p.o. Tag 4-21
* Pegfilgrastim 6 mg s.c day 8

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed AML defined according to the World Health Organization (WHO)-classification (excluding acute promyelocytic leukemia [APL])
* Ages 18-60 years
* Written informed consent of each patient at study entry.
* Molecular and cytogenetical diagnostics on initial bone marrow and peripheral blood specimen at the central reference laboratories

Exclusion Criteria:

* Bleeding independent of the AML
* Acute promyelocytic leukemia
* Uncontrollable infection
* Participation in a concurrent clinical study
* Insufficiency of the kidneys (creatinine > 1.5x upper normal serum level), of the liver (bilirubin, AST or AP > 2x upper normal serum level), severe obstructive or restrictive ventilation disorder, heart failure New York Heart Association (NYHA) III/IV
* Severe neurological or psychiatric disorder interfering with ability to give an informed consent.
* No consent for registration, storage and processing of the individual disease-characteristics and course.
* Performance status WHO > 2
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 920 (Actual)
Dates: Start 2004-07; Primary Completion 2011-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Complete remission (CR)-rate after induction therapy | after the second induction cycle
Relapse-free survival, one year after consolidation therapy with high-dose cytarabine considering different temporal sequences (1-3-5 versus 1-2-3) of the consolidation therapy | One year after consolidation therapy
Event-free survival | two years

SECONDARY OUTCOMES:
Kind, incidence, severity, temporal sequence and correlation of side effects of the study-drugs | during therapy
Cumulative incidence of relapse | two years
Cumulative incidence of death | two years
Overall survival | two years
Hematological recovery as well as incidence and duration of infections during neutropenia after each consolidation cycle | during consolidation therapy
Timely sequence of the pegfilgrastim-concentration in correlation to the absolute neutrophil counts after each consolidation cycle | during consolidation therapy
Hematologic and non-hematologic toxicity after consolidation therapy with high-dose cytarabine considering the different consolidation schemes (day 1-3-5 versus day 1-2-3) | during consolidation therapy
Days in hospital after each consolidation cycle | after consolidation therapy

CONTACTS AND LOCATIONS:
Overall Officials: Richard F Schlenk, Dr., Principal Investigator — University of Ulm
Locations (34):
- Austria (4):
  - Department of Hematology/Oncology, University Hospital Innsbruck, Innsbruck
  - Department of Internal Medicine I, Krankenhaus der Barmherzigen Schwestern, Linz
  - Medical Department III, St. Johann-Hospital, Salzburg
  - Center of Hematology and Oncology, Hanusch-Hospital, Vienna
- Germany (30):
  - Department of General Internal Medicine, University Hospital of Bonn, Bonn
  - Medical Department I, Hospital Bremen-Mitte, Bremen
  - Clinical Center of Hematology and Oncology, University Hospital of Düsseldorf, Düsseldorf
  - Department of Hematology and Oncology, Hospital Essen Süd, Ev. Hospital of Essen-Werden, Essen
  - Medical Department III, Hematology/Oncology, University of Frankfurt, Frankfurt
  - Department of Internal Medicine III, City Hospital Frankfurt am Main - Höchst, Frankfurt
  - Internal Medicine I, University of Freiburg, Freiburg im Breisgau
  - Medical Department IV, University Hospital of Giessen, Giessen
  - Department of Internal Medicine, Wilhelm-Anton-Hospital gGmbH, Goch
  - Centre of Internal Medicine, University Hospital Göttingen, Göttingen
  - Department of Oncology and Hematology, University Hospital Eppendorf, Hamburg
  - Medical Department II, Hematology and Oncology, General Hospital Altona, Hamburg
  - Medical Department III, Clinical Center Hanau, Hanau
  - Medical Department III, Hospital Hannover-Siloah, Hanover
  - Department of Hematology, Hematology and Oncology, Medizinische Hochschule Hannover, Hanover
  - Department of Internal Medicine I, University Hospital of Saarland, Homburg
  - Medical Department II, City Hospital Karlsruhe gGmbH, Karlsruhe
  - Medical Department II, University Hospital of Kiel, Kiel
  - Department of Internal Medicine/Hematology and Oncology, Cartias Hospital Lebach, Lebach
  - Department of Hematology and Oncology, Hospital of Lüdenscheid, Lüdenscheid
  - Department of Hematology and Internal Oncology, University Hospital of Mainz, Mainz
  - Medical Department III, Clinical Center Rechts der Isar, München
  - Department of Hematology and Oncology, Clinical Center of Oldenburg gGmbH, Oldenburg
  - Department of Hematology and Oncology, Caritas Hospital St. Theresia, Saarbrücken
  - Department of Oncology, Clinical Center of Stuttgart, Stuttgart
  - Medical Department II, Diakonie Hospital, Stuttgart
  - Medical Department I, Hospital of Barmherzige Brüder, Trier
  - Department of Internal Medicine II, University Hospital of Tübingen, Tübingen
  - Medical Clinic II-Hematology/Oncology, Hospital Villingen-Schwenningen, Villingen-Schwenningen
  - Medical Department I, Helios Hospital Wuppertal, Wuppertal

REFERENCES:
- [Result] Schlenk RF, Lubbert M, Benner A, Lamparter A, Krauter J, Herr W, Martin H, Salih HR, Kundgen A, Horst HA, Brossart P, Gotze K, Nachbaur D, Wattad M, Kohne CH, Fiedler W, Bentz M, Wulf G, Held G, Hertenstein B, Salwender H, Gaidzik VI, Schlegelberger B, Weber D, Dohner K, Ganser A, Dohner H; German-Austrian Acute Myeloid Leukemia Study Group. All-trans retinoic acid as adjunct to intensive treatment in younger adult patients with acute myeloid leukemia: results of the randomized AMLSG 07-04 study. Ann Hematol. 2016 Dec;95(12):1931-1942. doi: 10.1007/s00277-016-2810-z. Epub 2016 Oct 3. PMID 27696203
- [Derived] Schlenk RF, Kayser S, Bullinger L, Kobbe G, Casper J, Ringhoffer M, Held G, Brossart P, Lubbert M, Salih HR, Kindler T, Horst HA, Wulf G, Nachbaur D, Gotze K, Lamparter A, Paschka P, Gaidzik VI, Teleanu V, Spath D, Benner A, Krauter J, Ganser A, Dohner H, Dohner K; German-Austrian AML Study Group. Differential impact of allelic ratio and insertion site in FLT3-ITD-positive AML with respect to allogeneic transplantation. Blood. 2014 Nov 27;124(23):3441-9. doi: 10.1182/blood-2014-05-578070. Epub 2014 Sep 30. PMID 25270908
- [Derived] Gaidzik VI, Bullinger L, Schlenk RF, Zimmermann AS, Rock J, Paschka P, Corbacioglu A, Krauter J, Schlegelberger B, Ganser A, Spath D, Kundgen A, Schmidt-Wolf IG, Gotze K, Nachbaur D, Pfreundschuh M, Horst HA, Dohner H, Dohner K. RUNX1 mutations in acute myeloid leukemia: results from a comprehensive genetic and clinical analysis from the AML study group. J Clin Oncol. 2011 Apr 1;29(10):1364-72. doi: 10.1200/JCO.2010.30.7926. Epub 2011 Feb 22. PMID 21343560
- [Derived] Kayser S, Schlenk RF, Londono MC, Breitenbuecher F, Wittke K, Du J, Groner S, Spath D, Krauter J, Ganser A, Dohner H, Fischer T, Dohner K; German-Austrian AML Study Group (AMLSG). Insertion of FLT3 internal tandem duplication in the tyrosine kinase domain-1 is associated with resistance to chemotherapy and inferior outcome. Blood. 2009 Sep 17;114(12):2386-92. doi: 10.1182/blood-2009-03-209999. Epub 2009 Jul 14. PMID 19602710
- [Derived] Schlenk RF, Dohner K, Kneba M, Gotze K, Hartmann F, Del Valle F, Kirchen H, Koller E, Fischer JT, Bullinger L, Habdank M, Spath D, Groner S, Krebs B, Kayser S, Corbacioglu A, Anhalt A, Benner A, Frohling S, Dohner H; German-Austrian AML Study Group (AMLSG). Gene mutations and response to treatment with all-trans retinoic acid in elderly patients with acute myeloid leukemia. Results from the AMLSG Trial AML HD98B. Haematologica. 2009 Jan;94(1):54-60. doi: 10.3324/haematol.13378. Epub 2008 Dec 4. PMID 19059939